CLINICAL TRIAL: NCT06446531
Title: Pioneering and Affordable Strategies to Prevent Progression of Prediabetes, Obesity and CV Risk in Hispanics
Brief Title: Prevention of Progression of Prediabetes, Obesity and CV Risk
Acronym: Pre-DM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Baptist Health Foundation of San Antonio (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000485 Pre-DM
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Pre-Diabetes; Weight, Body; Cardiovascular Diseases
Keywords: Affordable strategies; Prevention of progression; Hispanic
MeSH Terms: conditions — Glucose Intolerance; Body Weight; Cardiovascular Diseases | interventions — semaglutide; empagliflozin; Tablets; Metformin; Pioglitazone

STUDY DESIGN:
Intervention Model Description: Single-blind Randomized, placebo-controlled trial.
Who Masked: Participant
Masking Description: This will be single blind study, given all treatment arms being pills, once subjects are randomized, they will not be told which mediation they are taking, and treatment will be dispensed in unmarked bottles at each timepoint.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Randomization will occur 1:1:1:1 to this placebo group
  Interventions: Drug: Placebo
- SGLT2 inhibitor Group (Experimental): Randomization will occur 1:1:1:1 to this SGLT2 inhibitor group
  Interventions: Drug: Jardiance 25Mg Tablet
- GLP-1 Receptor Agonist Group (Experimental): Randomization will occur 1:1:1:1 to this GLP-1 receptor agonist group
  Interventions: Drug: Rybelsus Tablet
- Metformin with SGLT2 Inhibitor Group (Experimental): Randomization will occur 1:1:1:1 to this metformin plus SGLT2 inhibitor group
  Interventions: Drug: Metformin; Drug: Actos

INTERVENTIONS:
Drug: Placebo — Oral tablet administered once daily
  Other Names: Zebbo
  Arms: Placebo
Drug: Rybelsus Tablet — Oral tablet started at a 3mg dose once daily and increased to 7mg once daily or maximum tolerable dose.
  Other Names: Semaglutide
  Arms: GLP-1 Receptor Agonist Group
Drug: Jardiance 25Mg Tablet — Oral 25 mg Sodium-Glucose Co-Transporter (SGLT2) inhibitor administered once daily
  Other Names: Empagliflozin
  Arms: SGLT2 inhibitor Group
Drug: Metformin — Oral tablet started at a dose of 500mg with an increase of 500mg weekly up to a maximum dose of 2000mg (4 tablets)
  Other Names: Metformin Hydrochloride
  Arms: Metformin with SGLT2 Inhibitor Group
Drug: Actos — Oral tablet dosed at 15mg once daily
  Other Names: Pioglitazone
  Arms: Metformin with SGLT2 Inhibitor Group

SUMMARY:
The investigators are studying how to help people with prediabetes (Pre-DM) and obesity. The goal is to use new and affordable treatments to bring blood sugar levels back to normal and help participants to lose weight. The investigators also want to reduce participants risk of heart problems. The study team will look at how these treatments affect metabolism and other body functions to help find new ways to treat diabetes and obesity in the future.

DETAILED DESCRIPTION:
While taking part in this study, participants will be asked to attend approximately 16 visits with the researchers or study staff.

Study participants are assigned (single-blinded, only the study team will know the assigned group) to one of 4 study groups, receiving a 6-month treatment with Nutritional Consultation + either SGLT2 Inhibitor (Empagliflozin), Rybelsus (GLP1 Receptor Agonist), Metformin + Pioglitazone, or placebo. A placebo is an inactive, harmless substance that looks like the other study drugs. This study does not require overnight stays at the hospital in any of the study groups.

Duration of the Study will be about 6-7 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will have an established diagnosis of pre-Diabetes Mellitus (DM) before the screening visit, documented by an acceptable modality in the last 6 months.
2. Age ≥ 18 years old
3. Body Mass Index (BMI)=25-40 kg/m2
4. Glycated Hemoglobin (HbA1c) = 5.7-6.4%
5. Blood Pressure (BP) <160/100
6. Estimated Glomerular Filtration Rate (eGFR) ≥30 ml/min•1.73m2
7. Body weight must be stable (±5 pounds) over the last 3 months.
8. Oral diuretics, if prescribed to the patient according to local guidelines and discretion of the investigator, should be stable for at least 1 week prior to randomization.
9. Hispanic ethic group
10. Willing to adhere to medication regimen for up to 6 months.
11. Male or female, if female, met these criteria:

    1. Not pregnant or breast-feeding
    2. Negative pregnancy test result at visit 1 (screening)
    3. During the entire study, women of childbearing potential (WOCBP) including peri-menopausal women who have a menstrual period within 1 year must practice appropriate, and effective birth control, either implants or pills, or a vasectomized partner prior to receiving the first dose of study medication
12. Does not suffer from severe claustrophobia
13. No contraindication for Magnetic Resonance Imaging (MRI) (metal plates, screws, shrapnel, pins, or cardiac pacemaker)

Exclusion Criteria:

1. Patients currently on one of the selected therapies
2. Extended diagnoses with Type 2 Diabetes
3. Pregnancy, lactation, women of childbearing age (WOCBA) unwilling to use contraception
4. Known allergy/sensitivity to study drugs or their ingredients
5. Major oncologic diagnosis in the last 5 years
6. Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
7. Inability or unwillingness of individual or legal guardian/representative to give written informed consent
8. Major organ or metabolic diseases, or physical limitations that will not allow the subject to complete the study
9. Myocardial infraction, coronary artery bypass graft surgery, or other major cardiovascular event in the past 60 days
10. Heart transplant recipient or listed for a heart transplant
11. Currently implanted left ventricular assist device
12. Cardiomyopathy based on infiltrative or cumulative hypertrophic obstructive cardiomyopathy or known pericardial constriction
13. Any severe (obstructive or regurgitant) valvular heart disease, expected to lead to surgery during the trial period
14. Acute decompensated heart failure requiring intravenous diuretics, vasodilators, inotropic agents, or mechanical support within 1 week of screening and during the screening period prior to randomization
15. Implanted cardioverter defibrillator within 3 months prior to screening
16. Cardiac resynchronization therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c Level (HBA1c) | Baseline and 6 months
  Percentage of glycated hemoglobin level in blood

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Baseline and 6 months
  Measure of body fat based on height and weight that applies to adult men and women
Percentage of Body Fat Composition | Baseline and 6 months
  Measurement of body fat using a DEXA scan
Left Ventricular Function | Baseline and 6 months
  Cardiac function is measured by left-ventricular function measured using cardiac MRI and expressed as a percentage
Measure of phosphocreatine k-value | Baseline and 6 months
  A skeletal muscle bioenergetic measurement using skeletal muscle MRI/MRS
Measure of oxidative capacity | Baseline and 6 months
  A skeletal muscle bioenergetic measurement using skeletal muscle MRI/MRS
Measure of intramyocellular lipids (IMCL) | Baseline and 6 months
  A skeletal muscle bioenergetic measurement using skeletal muscle MRI/MRS
Measure of extramyocellular lipids (EMCL) | Baseline and 6 months
  A skeletal muscle bioenergetic measurement using skeletal muscle MRI/MRS
Patient Reported Outcomes (PROMIS) | Baseline and 6 months
  A survey used to assess physical function. Subjects will rank 20 questions from a scale of 1 - 5, with 5 being the highest physical function and 1 being the lowest. The score will be added up, and the Raw score will be converted to T-Score using the PROMIS Adult v2.0 Physical Function 20a Short Form Conversion Table. The range of T-scores is 12.1-62.5. A higher score indicates higher physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Solis-Herrera, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The Institution or respective designees may present or publish the results of a scientific investigation involving this Study in accordance with International Committee of Medical Journal Editors (ICMJE). The Sponsor Investigator, funding agency, or PI initiating the study will collaborate to determine who has publication rights for authorship upon review and approval of proposed manuscripts.
Supporting Information: Study Protocol, SAP
Time Frame: At the time of publication in a peer review journal